CLINICAL TRIAL: NCT02032498
Title: Evaluation of Near- InfraRed Imaging of ICG in Comparison With the Lymphoscintigraphic Technique Using Intramammary and Peritumoral Injection of 99mTc-HSA-Nanocolloids for the SLN Detection in BC Patients.
Brief Title: Evaluation of Two Techniques for the SLN Detection in BC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-001555-12
Record Dates: First submitted 2013-11-20; First posted 2014-01-10 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
Keywords: sentinel lymph nodes; radiocolloids; Indocyanine Green; complementarity; axillary lymph node dissection
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Indocyanine Green (Experimental): superficial injections of Indocyanine Green in the breast
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Superficial injection of ICG in combination with deep injection of 99mTc-HSA to evaluate the complementarity of the two techniques
  Other Names: ICG

SUMMARY:
The revision of our data shows that since its introduction in our institution (Jules Bordet Institute) in 1998 (until 2010, the year of the last review of cases), 53 patients underwent neoadjuvant therapy before selective sentinel lymph node dissection followed by conventional axillary dissection.

The analysis of these cases shows that:

* The lack of demonstration of sentinel lymph nodes observed in 8 cases (6 cN0) is associated in 75% of them with a pN+ status
* If scintigraphic imaging is "positive" (demonstration of the sentinel lymph nodes: 35 cN0 and 10 cN+), our results appear favorable with a single false negative SLN result (False Negative Rate = 1/20 or 5%).

Therefore we propose additional technique for LN detection by indocyanine green, we hypothesize that the combination of two different injections improves the technique of sentinel lymph node biopsy.

DETAILED DESCRIPTION:
The principal objective of this study is to evaluate the detection rate, the false negative rate and the overall accuracy of the lymphofluoroscopic research of the sentinel lymph nodes after periareolar injections of Indocyanine Green (ICG) in combination and in comparison with our classical intramammary and peritumoral injections of 99mTc-HSA-Nanocolloids in patients with breast cancer. These patients are currently out of the inclusion criteria and still undergo systematically complete axillary node dissection.

In this study (which would include at least 200 patients over a period of 2 years, with at least 100 patients after neoadjuvant chemotherapy) the involved surgeons would continue to perform complete axillary node dissections.

The radioactive SLN would be retrieved ex vivo in the axillary piece (with the gamma probe, after intramammary and peritumoral injections of radiocolloids the day before the surgery, or at least 3 hours before, with scintigraphic preoperative images as already performed routinely for patients described in the introduction 1 of this letter). These radioactive lymph nodes would thereafter been controlled for their possible fluorescence (with our fluorescence camera and after periareolar injection of ICG in the operating room just before the surgery). Finally, in the service of Pathology, all the lymph nodes found by the pathologist in the axillary piece will be controlled for their possible fluorescence.

With this approach, the surgeon will not have to search for SLN and the operative duration will not be extended.

Secondary objectives:

The current literature about the results of SLNB technique has not yet considered the influence of the addition of SPECT-CT imaging (standard approach in our institute since more than 3 years) to planar imaging. In this study, we propose to analyse in a prospective manner the contribution of SPECT-CT: contribution of the analysis of the signal intensity of active lymph nodes on SPECT slides to define a resection threshold corresponding to lymph nodes at risk of being pN+, accuracy for the anatomic localization, better accuracy of the number of SLN on the SPECT-CT versus planar image, better definition of the number of lymph nodes (to be analysed on the CT) covered by a radioactive spot (we have already observed 3 adjacent lymph nodes under one only active spot).

In this last case, such spots covering several lymph nodes would be analysed for the possible fluorescence of each lymph node.

The fluorescence of the detected lymph nodes will be analysed semi-quantitatively and related to their pN+ characteristics (pNi, pNµ, pN1, pNmacro). This first analysis may have major implications when our surgeons will perform an in vivo research of fluorescent SLN (see also Bourgeois et al. 2003).

Finally, we propose to analyse the kinetic and the vascular characteristics (aspects of the vessels on the images) of ICG migration from its injection point to the axilla. We will try to define possible predictive parameters of extended and/or macroscopic involvement of axillary lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Female patients submitted to mastectomy or tumorectomy with Complete Axillary Node Dissection (but to whose SLN procedure might be proposed in the future).
* General operability.
* Informed consent form signed

Exclusion Criteria:

* Age less than18 years old.
* Former operation in the axilla and/or breast.
* Any previous radiotherapy at the concerned breast and/or axilla and/or chest wall.
* History of allergy or hypersensitivity against the investigational product (its active substance or ingredients), to iodine or to shellfish.
* Apparent hyperthyroidism, autonomous thyroid adenoma, unifocal, multifocal or disseminated autonomies of the thyroid gland.
* Documented coronary disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
false negative rate for each technique (fluorescence and radiocolloids) | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Nogaret, MD, Principal Investigator — Surgeon
Locations (1):
- Jules Bordet Institute, Brussels, Brussels Capital, Belgium